CLINICAL TRIAL: NCT03298659
Title: Instantaneous Wave-free Ratio Guided Multi-vessel revascularizatiOn During Percutaneous Coronary intervEntion for Acute myocaRdial iNfarction (iMODERN)
Brief Title: iFR Guided Multi-vessel Revascularization During Percutaneous Coronary Intervention for Acute Myocardial Infarction
Acronym: iMODERN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Volcano Europe BVBA/SPRL (Unknown); Biotronik AG (Industry); Stichting Life Sciences & Health (Unknown); Duke Cardiovascular Magnetic Resonance Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL60107.029.16
Record Dates: First submitted 2017-09-18; First posted 2017-10-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction; Multi Vessel Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to (A) an active treatment arm with complete, iFR-guided revascularization of every noninfarct coronary lesion >50% and iFR ≤0.89; or (B) a deferred treatment arm, in which patients will undergo an adenosine stress perfusion CMR scan within 6 weeks after STEMI, with revascularization of the noninfarct coronary lesions with associated perfusion defects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active iFR-guided revascularization (Experimental): Decision to treat the nonculprit coronary stenosis if there is a significant pressure drop over the stenosis, as measured by intracoronary iFR assessment
  Interventions: Diagnostic Test: iFR
- Deferred CMR-guided revascularization (Active Comparator): Decision to treat the nonculprit coronary stenosis if perfusion defect visible in corresponding coronary territory as visualized on stress perfusion CMR imaging
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: iFR — Treatment guided by instantaneous wave-free ratio
  Arms: Active iFR-guided revascularization
Diagnostic Test: CMR — Treatment guided by stress perfusion CMR
  Arms: Deferred CMR-guided revascularization

SUMMARY:
In patients with acute ST-elevation myocardial infarction (STEMI), 40-60% have multi-vessel disease with an increased cardiovascular morbidity and mortality. Although it is not recommended to revascularize noninfarct lesions during the acute intervention, recent investigations suggest the opposite and show improved outcome after direct revascularization of noninfarct lesions. It is undesirable to risk procedure-related complications by treating noninfarct lesions without impaired flow. It is currently unknown whether pressure guided revascularization of noninfarct lesions in the acute phase improves outcome compared to the current guidelines.

The iMODERN trial aims to compare an iFR-guided intervention of noninfarct lesions during the acute intervention with a deferred stress perfusion CMR-guided strategy during the outpatient follow-up, to determine the optimal therapeutic approach for STEMI patients with multivessel lesions.

DETAILED DESCRIPTION:
Study design:

The study is a prospective, randomized controlled, multicentre study.

Study population:

The research population will be recruited from the general patient population presenting with an acute STEMI. Patients treated with successful primary PCI and one or more additional significant coronary lesions in another coronary artery will be enrolled in the study. A total of 1,146 consecutive patients will be included.

Intervention:

The patients will be randomized 1:1, to (A) an active treatment arm with complete, iFR-guided revascularization of every noninfarct coronary lesion >50% and iFR ≤0.89; (B) a deferred treatment arm, in which patients will undergo an adenosine stress perfusion CMR scan within 6 weeks after STEMI, with revascularization of the noninfarct coronary lesions with associated perfusion defects.

Main study parameters/endpoints:

The primary end point consists of a combined outcome, including all-cause death, recurrent MI and hospitalization for heart failure at 3 years follow-up.

Duration:

Anticipated recruitment is 2 years. Follow-up will be performed at 6 months, 12 months, 3 years and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinical presentation of STEMI and successful primary PCI within 12 hours from onset of symptoms.
* One or more other, noninfarct coronary artery lesions of >50% stenosis and feasible to be revascularized (i.e. minimal diameter 2mm).

Exclusion Criteria:

* History of myocardial infarction.
* Hemodynamic instability, respiratory failure, Kilips class ≥III.
* Known GFR<30 ml/min.
* Known contra-indications for stress CMR (e.g.: severe claustrophobia, metal implants, severe renal failure, severe astma).
* Refusal or inability to provide informed consent.
* Life expectancy due to noncardiovascular co-morbidity of less than 12 months.
* Chronic total occlusion.
* Left main stem stenosis (>50%).
* Residual noninfarct lesion in infarct coronary artery.
* Complex (e.g. bifurcation) noninfarct target lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1146 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite end point of Major Adverse Cardiac Events | 3 years
  All-cause death, recurrent myocardial infarction and hospitalization for heart failure

SECONDARY OUTCOMES:
All cause mortality | 6 and 12 months, 3 and 5 years
  All cause mortality at 6 and 12 months, 3 and 5 years
Cardiovascular mortality | 6 and 12 months, 3 and 5 years
  Cardiovascular mortality at 6 and 12 months, 3 and 5 years
Myocardial infarction | 6 and 12 months, 3 and 5 years
  Myocardial infarction at 6 and 12 months, 3 and 5 years
Cerebral events | 6 and 12 months, 3 and 5 years
  Stroke and transient ischemic attack
Major bleeding | 6 months
  Haemorrhagic complications
Unstable angina | 6 and 12 months, 3 and 5 years
  Unstable angina including ECG-changes at 6 and 12 months, 3 and 5 years
Coronary angiography | 6 and 12 months, 3 and 5 years
  Coronary angiography at 6 and 12 months, 3 and 5 years
Revascularization | 6 and 12 months, 3 and 5 years
  Any revascularization at 6 and 12 months, 3 and 5 years
Target lesion failure | 6 and 12 months, 3 and 5 years
  Failure and/or revascularization by percutaneous or surgical methods of the target lesion
Stent thrombosis | 6 and 12 months, 3 and 5 years
  Stent thrombosis at 6 and 12 months, 3 and 5 years
Cost effectiveness analysis | 6 and 12 months, 3 and 5 years
  Costs related to complete, iFR-guided revascularization versus CMR-guided treatment, including cost utility analysisfrom a societal perspective with the costs per prevented cardiac eventand the costs per QALY as the respective primary health economic outcomes (using a quality of life questionnaire and a health care resource use questionnaire)
Quality of life | 6 and 12 months, 3 and 5 years
  Quality of life questionnaires, i.e. SAQ, EQ-5D-5L and Minnesota heart failure questionnaire, at 6 and 12 months, 3 and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nijveldt R, Maeng M, Beijnink CWH, Piek JJ, Al-Lamee RK, Raposo L, Baptista SB, Escaned J, Davies J, Klem I, Yosofi B, van Geuns RM, Frederiksen CA, Jakobsen L, El Barzouhi A, van der Heijden DJ, Ilhan M, Rasoul S, Brinckman S, Saraber C, Jones DA, Petersen SE, Podlesnikar T, Bunc M, Beijk MAM, Piers LH, van Rees JB, Seligman H, Cole G, Iglesias JF, Degrauwe S, van 't Hof AWJ, Lipsic E, Pundziute-do Prado G, Chattranukulchai P, Rodriguez-Palomares JF, Rigger J, Meuwissen M, Kleijn L, Pereira B, Monti L, van der Schaaf RJ, Sanchis J, Belli G, Tijssen JGP, Thim T, van Royen N; iMODERN Investigators. Immediate or Deferred Nonculprit-Lesion PCI in Myocardial Infarction. N Engl J Med. 2025 Oct 28. doi: 10.1056/NEJMoa2512918. Online ahead of print. PMID 41159879
- [Derived] Ong P, Martinez Pereyra V, Sechtem U, Bekeredjian R. Management of patients with ST-segment myocardial infarction and multivessel disease: what are the options in 2022? Coron Artery Dis. 2022 Sep 1;33(6):485-489. doi: 10.1097/MCA.0000000000001157. Epub 2022 Jul 11. PMID 35811565
- [Derived] Beijnink CWH, Thim T, van der Heijden DJ, Klem I, Al-Lamee R, Vos JL, Koop Y, Dijkgraaf MGW, Beijk MAM, Kim RJ, Davies J, Raposo L, Baptista SB, Escaned J, Piek JJ, Maeng M, van Royen N, Nijveldt R. Instantaneous wave-free ratio guided multivessel revascularisation during percutaneous coronary intervention for acute myocardial infarction: study protocol of the randomised controlled iMODERN trial. BMJ Open. 2021 Jan 15;11(1):e044035. doi: 10.1136/bmjopen-2020-044035. PMID 33452200